CLINICAL TRIAL: NCT04273828
Title: Impact of Muscle Degeneration in Chronic Ow Back Pain in Patients Undergoing Neural Decompression
Brief Title: Impact of Muscle Degeneration in Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: 94868618.7.0000.0071
Record Dates: First submitted 2020-02-11; First posted 2020-02-18 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-11

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Radiculopathy; Back Pain
Keywords: back pain; lumbar disc herniation; lumbar spinal stenosis; Decompression, surgical
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Radiculopathy; Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Lumbar decompressive surgery — Patients with lumbar degenerative diseases and symptoms of nerve compression (radiculopathy or neurogenic claudication) who will undergo surgical treatment for neural decompression (discectomy, foraminotomy or laminectomy).

SUMMARY:
Surgical interventions for the removal of intervertebral disc fragments or to enlarge a narrow spine canal are commonly performed worldwide and are considered efficient. Concomitant low back pain is not uncommon among patients with lumbar nerve compression and neurological symptoms. When present, controversy persists in the literature regarding its ideal management. Although neurological symptoms improve after decompressive surgery, the presence of residual chronic low back pain may worsen satisfaction scores and cause functional disability.

The hypothesis of the present study is that the presence of atrophy of the paraspinal and trunk muscles predicts chronic low back pain after lumbar neural decompression. If confirmed, this finding will aid in better planning of physical rehabilitation strategies for this group of patients, as well as a clearer prediction regarding surgical treatment outcomes for patients and health professionals.

DETAILED DESCRIPTION:
This is a prospective cohort study. Patients with lumbar degenerative diseases and symptoms of nerve compression (radiculopathy or neurogenic claudication) who will undergo surgical treatment for neural decompression (discectomy, foraminotomy or laminectomy).

The cohort will be followed by a team researcher (not blinded to the purpose of the study) at preoperative (up to 1 month before surgery), immediate postoperative (12 to 24 hours after procedure), 06, 12 and 24 months after surgery. Imaging tests will be performed on the preoperative evaluation and at six months follow-up after the operation.

The treatment will consist of lumbar decompression surgery, which may consist of discectomy, foraminotomy or laminectomy, according to the type and location of the compression. The choice of surgical technique will be made by the assistant surgeon.

Patients will be divided into four groups regarding the type of soft tissue retractor and image magnification:

Group 1: (minimally invasive microdiscectomy): surgeries performed with loupes or microscope plus minimally invasive soft tissue retractors (tubular or "Caspar").

Group 2: (open microdiscectomy) surgeries performed with loupes or microscope plus conventional soft tissue retractors (auto static, "Taylor" or "McCulloch").

Group 3: (endoscopic discectomy): surgeries performed by means of the "full endoscopic" technique;

Group 4: (open discectomy "with the naked eye"): surgeries performed without image magnification. Use of conventional soft tissue retractors (auto static, "Taylor" or "McCulloch").

Image Evaluation:

1. X-Rays (anteroposterior, lateral, dynamic lateral films) - to evaluate and measure the presence of scoliosis, spondylolisthesis or Degenerative vertebral dislocations.
2. MRI: to detect and to grade the presence of fat infiltration of the Psoas and Multifidus muscles (Arabanas et al); to grade Modic Signal and facet joint degeneration (Weishaupt et al).

Sample size:

For the sample size estimation, we considered the main outcome of the study, a 1.5-point change in the pain scale (VAS) among patients with fat infiltration (grades 1, 2, or 3) and without fat infiltration (grade 0), after 6 months of spine surgery, with 80% power and 95% confidence, the sample required for the study is 28 patients in each group considering a two-tailed test. Similarly to the previous study, we observed that the first 14 patients in the pilot study, 20% of patients had without fat infiltration, therefore, as the admission of patients into the study is consecutive, we expect to find this same percentage of patients without fat infiltration in the final sample of patients, so 140 patients are needed to get 28 patients without fat infiltration. Predicting a loss of 20% of patients at 6 months of follow-up, the initial sample to be considered will be 168 patients to obtain the minimum number of patients required in each group.

Statistics:

Numerical variables with normal distribution will be described by means and standard deviations and variables with non-normal distribution by medians and interquartile ranges, in addition to the minimum and maximum values. The distributions of numerical variables will be verified by histograms, boxplots, and, if necessary, Shapiro-Wilk normality tests. Categorical variables will be described by absolute frequencies and percentages. The analyzes will be performed with the SPSS26 program, considering a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

1. adults 18 years of age and older;
2. with symptoms of lumbosacral neural compression (radiculopathy or neurogenic lameness);
3. failed conservative treatment for at least 6 weeks;
4. undergoing surgery for neural decompression (discectomy and / or foraminotomy and / or hemilaminectomy);
5. with complete pre and postoperative medical records in all evaluations.

Exclusion Criteria:

1. need for lumbar arthrodesis;
2. deep infection requiring surgical cleaning;
3. patients submitted to joint facet rhizotomy;
4. active rheumatologic disease, including seronegative arthropathies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at the Israelita Albert Einstein Hospital (HIAE), a tertiary private philanthropic hospital located in the city of São Paulo, Brazil. All participants will be from and treated at the institution's spine surgery outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity | Baseline, 3, 6, 12 and 24 months after surgery
  Pain intensity will be measured using VAS 0-10 (0 being no pain and 10 maximum pain)

SECONDARY OUTCOMES:
Radiological evaluation | Baseline and 6 month after surgery
  Magnetic resonance imaging (MRI) reading parameters of Paravertebral and Psoas major fat tissue infiltration follow the standardized institutional protocol for spine evaluation.
Change in Kinesiophobia | Baseline, 3, 6, 12 and 24 months after surgery
  Assessment of fear avoidance beliefs related to physical activity and work will be evaluated by the questionnaire Fear avoidance Beliefs Questionnaire (FABQ)
Change in Psychosocial Risk Prognosis | Baseline, 3, 6, 12 and 24 months after surgery
  Psychosocial risk prognosis will be measured by the brazilian version of the STarT Back screening tool.
Change in Global Impression of Recovery | Baseline, 3, 6, 12 and 24 months after surgery
  Global impression of recovery will be measured by the Global Perceived Effect of Change(GPE)
Change in Mood Disorders in The setting of Medical Practice | Baseline, 3, 6, 12 and 24 months after surgery
  Anxiety and depression aspects will be measured by the Hospital Anxiety and Depression Scale (HADS)
Change in Disability | Baseline, 3, 6, 12 and 24 months after surgery
  Disability will be measured by the Oswestry Disability Index, Brazilian version 2.0.
Change in Quality life | Baseline, 3, 6, 12 and 24 months after surgery
  EuroQoL will be combined with a Visual Analogue Scale(VAS) to carry out the cost-effectiveness analysis of the second opinion program.

OTHER OUTCOMES:
Sociodemographic characteristics | Baseline
  Age (years), sex (male or female), body mass index (BMI), formal education (years of study), type of occupation (carrying weight or not).

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Gotfryd, PhD, Principal Investigator — Phisician
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bae HW, Rajaee SS, Kanim LE. Nationwide trends in the surgical management of lumbar spinal stenosis. Spine (Phila Pa 1976). 2013 May 15;38(11):916-26. doi: 10.1097/BRS.0b013e3182833e7c. PMID 23324922
- [Background] Kovacs FM, Urrutia G, Alarcon JD. Surgery versus conservative treatment for symptomatic lumbar spinal stenosis: a systematic review of randomized controlled trials. Spine (Phila Pa 1976). 2011 Sep 15;36(20):E1335-51. doi: 10.1097/BRS.0b013e31820c97b1. PMID 21311394
- [Background] Jacobs WC, van Tulder M, Arts M, Rubinstein SM, van Middelkoop M, Ostelo R, Verhagen A, Koes B, Peul WC. Surgery versus conservative management of sciatica due to a lumbar herniated disc: a systematic review. Eur Spine J. 2011 Apr;20(4):513-22. doi: 10.1007/s00586-010-1603-7. Epub 2010 Oct 15. PMID 20949289
- [Background] Bydon M, De la Garza-Ramos R, Macki M, Baker A, Gokaslan AK, Bydon A. Lumbar fusion versus nonoperative management for treatment of discogenic low back pain: a systematic review and meta-analysis of randomized controlled trials. J Spinal Disord Tech. 2014 Jul;27(5):297-304. doi: 10.1097/BSD.0000000000000072. PMID 24346052
- [Background] Hansen L, de Zee M, Rasmussen J, Andersen TB, Wong C, Simonsen EB. Anatomy and biomechanics of the back muscles in the lumbar spine with reference to biomechanical modeling. Spine (Phila Pa 1976). 2006 Aug 1;31(17):1888-99. doi: 10.1097/01.brs.0000229232.66090.58. PMID 16924205
- [Background] Freeman MD, Woodham MA, Woodham AW. The role of the lumbar multifidus in chronic low back pain: a review. PM R. 2010 Feb;2(2):142-6; quiz 1 p following 167. doi: 10.1016/j.pmrj.2009.11.006. PMID 20193941
- [Background] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653
- [Background] Vigatto R, Alexandre NM, Correa Filho HR. Development of a Brazilian Portuguese version of the Oswestry Disability Index: cross-cultural adaptation, reliability, and validity. Spine (Phila Pa 1976). 2007 Feb 15;32(4):481-6. doi: 10.1097/01.brs.0000255075.11496.47. PMID 17304141
- [Background] 11. Herdman M, Fox-Rushby J, Rabin R, Badia X, Selai C. Producing other language versions of the EQ-5D. In: Brooks R, Rabin R, de Charro F (eds). The measurement and valuation of health status using EQ-5D: A European perspective. Kluwer Academic Publishers 2003.
- [Background] Abreu AM, Faria CD, Cardoso SM, Teixeira-Salmela LF. [The Brazilian version of the Fear Avoidance Beliefs Questionnaire]. Cad Saude Publica. 2008 Mar;24(3):615-23. doi: 10.1590/s0102-311x2008000300015. Portuguese. PMID 18327449
- [Background] Pilz B, Vasconcelos RA, Marcondes FB, Lodovichi SS, Mello W, Grossi DB. The Brazilian version of STarT Back Screening Tool - translation, cross-cultural adaptation and reliability. Braz J Phys Ther. 2014 Sep-Oct;18(5):453-61. doi: 10.1590/bjpt-rbf.2014.0028. Epub 2014 Aug 29. PMID 25372008
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Marcolino JA, Mathias LA, Piccinini Filho L, Guaratini AA, Suzuki FM, Alli LA. Hospital Anxiety and Depression Scale: a study on the validation of the criteria and reliability on preoperative patients. Rev Bras Anestesiol. 2007 Feb;57(1):52-62. doi: 10.1590/s0034-70942007000100006. English, Portuguese. PMID 19468618
- [Background] Arbanas J, Pavlovic I, Marijancic V, Vlahovic H, Starcevic-Klasan G, Peharec S, Bajek S, Miletic D, Malnar D. MRI features of the psoas major muscle in patients with low back pain. Eur Spine J. 2013 Sep;22(9):1965-71. doi: 10.1007/s00586-013-2749-x. Epub 2013 Mar 31. PMID 23543369
- [Background] Kjaer P, Bendix T, Sorensen JS, Korsholm L, Leboeuf-Yde C. Are MRI-defined fat infiltrations in the multifidus muscles associated with low back pain? BMC Med. 2007 Jan 25;5:2. doi: 10.1186/1741-7015-5-2. PMID 17254322
- [Background] Kader DF, Wardlaw D, Smith FW. Correlation between the MRI changes in the lumbar multifidus muscles and leg pain. Clin Radiol. 2000 Feb;55(2):145-9. doi: 10.1053/crad.1999.0340. PMID 10657162
- [Background] Ogawa M, Lester R, Akima H, Gorgey AS. Quantification of intermuscular and intramuscular adipose tissue using magnetic resonance imaging after neurodegenerative disorders. Neural Regen Res. 2017 Dec;12(12):2100-2105. doi: 10.4103/1673-5374.221170. PMID 29323052
- [Background] Modic MT, Steinberg PM, Ross JS, Masaryk TJ, Carter JR. Degenerative disk disease: assessment of changes in vertebral body marrow with MR imaging. Radiology. 1988 Jan;166(1 Pt 1):193-9. doi: 10.1148/radiology.166.1.3336678.
- [Background] Jarvinen J, Karppinen J, Niinimaki J, Haapea M, Gronblad M, Luoma K, Rinne E. Association between changes in lumbar Modic changes and low back symptoms over a two-year period. BMC Musculoskelet Disord. 2015 Apr 22;16:98. doi: 10.1186/s12891-015-0540-3. PMID 25897658
- [Background] Weishaupt D, Zanetti M, Boos N, Hodler J. MR imaging and CT in osteoarthritis of the lumbar facet joints. Skeletal Radiol. 1999 Apr;28(4):215-9. doi: 10.1007/s002560050503. PMID 10384992